CLINICAL TRIAL: NCT01860404
Title: Head Injury Treatment With Healthy and Advanced Dietary Supplements (HIT HEADS): A Randomized, Placebo-controlled, Double-blinded, Therapeutic Exploratory Clinical Trial of Branched Chain Amino Acids (BCAA's) in the Treatment of Concussion
Brief Title: BCAA Supplementation for Concussion
Acronym: HIT_HEADS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: The Dana Foundation (Other); Main Line Health (Other); University of Pennsylvania (Other); Pennsylvania Department of Health (Other Government)
Responsible Party: Principal Investigator, Sage R Myers, Attending Physician, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-010227
Record Dates: First submitted 2013-05-20; First posted 2013-05-22 (Estimated); Results first posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Brain Concussion
Keywords: Concussion; Branched chain amino acids; BCAA; HIT HEADS
MeSH Terms: conditions — Brain Concussion | interventions — Amino Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo will be administered orally twice daily for 21 days
  Interventions: Drug: Placebo solution
- Branched Chain Amino Acids (27g BID) (Experimental): 27 grams of BCAA's will be administered twice-daily for 21 days
  Interventions: Drug: Branched Chain Amino Acids
- Branched Chain Amino Acids (22.5g BID) (Experimental): 22.5 grams of BCAA's will be administered twice-daily for 21 days
  Interventions: Drug: Branched Chain Amino Acids
- Branched Chain Amino Acids (15g BID) (Experimental): 15 grams of BCAA's will be administered twice-daily for 21 days
  Interventions: Drug: Branched Chain Amino Acids
- Branched Chain Amino Acids (7.5g BID) (Experimental): 7.5 grams of BCAA's will be administered twice-daily for 21 days
  Interventions: Drug: Branched Chain Amino Acids

INTERVENTIONS:
Drug: Branched Chain Amino Acids — The three BCAA's will be combined together and dissolved in a flavored solution.
  Arms: Branched Chain Amino Acids (15g BID); Branched Chain Amino Acids (22.5g BID); Branched Chain Amino Acids (27g BID); Branched Chain Amino Acids (7.5g BID)
Drug: Placebo solution — The placebo solution will have similar taste, texture, consistency and appearance as the BCAA solution.
  Arms: Placebo

SUMMARY:
This study is a randomized, placebo-controlled, double-blinded, therapeutic exploratory clinical trial of branched chain amino acids (BCAA's) in the treatment of concussion. The aim of the study is to determine whether, compared to placebo treatment, administration of BCAA's, at one or more doses, after a concussion improves neurocognitive recovery at one or more time-periods post concussion.

DETAILED DESCRIPTION:
Annually, between 100,000 to 140,000 children present to the emergency department for concussion in the United States.1 The Centers for Disease Control now estimates that 1.6 - 3.8 million sports related concussions occur each year in the United States. A large proportion of these patients have enduring cognitive and neurobehavioral problems. Concussion is a heterogeneous insult to the brain that precipitates a complex pathophysiological process that can result in a cascade of deleterious side effects. At present, there are no proven therapies to mitigate or prevent the neurocognitive and neurobehavioral consequences of concussions. The limbic hippocampus, a brain structure crucial for learning and memory, is often damaged in concussion. In preclinical studies in our laboratory, analysis of ipsilateral hippocampi isolated from mice after traumatic brain injury (TBI) demonstrated that only the concentrations of the three BCAA's (valine, isoleucine, and leucine) were significantly altered (reduced) after injury. When these brain-injured animals received dietary supplementation with BCAA's, the concentrations of these amino acids were restored in the injured hippocampus and the injured animals demonstrated significant cognitive improvement to levels comparable to those obtained in non-injured control animals. In light of these results and the increasing awareness and morbidity associated with concussion, we are proposing a pilot therapeutic exploratory clinical trial to determine the effects of BCAA's in reducing the neurocognitive side effects of concussion injury.

ELIGIBILITY:
Inclusion Criteria

1. Males and females, ages 11 - 34 years, of any race.
2. Subjects who had a concussion, as diagnosed by a qualified physician, within 72 hours prior to enrollment.
3. Ability to have daily email and internet access.
4. Females must have a negative urine pregnancy test and must use an acceptable method of contraception.
5. Subjects must, in the opinion of the referring physician, have the capacity to provide informed consent.
6. Informed consent by the subject, or for subjects <18 years old both informed consent by a parent/guardian and child assent.

Exclusion Criteria

1. Witnessed seizure at the time of injury or penetrating head injury.
2. Prior concussion or TBI within 90 days.
3. Concussion or TBI severe enough to require admission to an intensive care unit for observation or intervention.
4. Previous history of TBI or concussion requiring admission to the hospital, disabling stroke, epilepsy, brain tumor, neurodegenerative condition, or psychiatric disease.
5. Subjects taking neurological or psychoactive medications as a regular daily prescription medication.
6. Known history of maple syrup urine disease or known family history of maple syrup urine disease.
7. Any investigational drug use within 30 days prior to enrollment.
8. Allergy to Food, Drug, and Cosmetic (FD&C) Red #40 (red dye 40) or Sucralose.
9. Lactating females.
10. Parents/guardians or subjects who, in the opinion of the investigators, may be non-compliant with study schedules or procedures.

Ages: 11 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2023-01 (Actual); Study Completion 2023-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sage Myers, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Cole JT, Mitala CM, Kundu S, Verma A, Elkind JA, Nissim I, Cohen AS. Dietary branched chain amino acids ameliorate injury-induced cognitive impairment. Proc Natl Acad Sci U S A. 2010 Jan 5;107(1):366-71. doi: 10.1073/pnas.0910280107. Epub 2009 Dec 7. PMID 19995960

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo will be administered orally twice daily for 21 days
  Placebo solution: The placebo solution will have similar taste, texture, consistency and appearance as the branched chain amino acid (BCAA) solution.
- Branched Chain Amino Acids (7.5g BID): 7.5 grams of BCAAs will be administered twice-daily for 21 days
  Branched Chain Amino Acids: The three BCAAs will be combined together and dissolved in a flavored solution.
- Branched Chain Amino Acids (15g BID): 15 grams of BCAAs will be administered twice-daily for 21 days
  Branched Chain Amino Acids: The three BCAA's will be combined together and dissolved in a flavored solution.
- Branched Chain Amino Acids (22.5g BID): 22.5 grams of BCAAs will be administered twice-daily for 21 days
  Branched Chain Amino Acids: The three BCAAs will be combined together and dissolved in a flavored solution.
- Branched Chain Amino Acids (27g BID): 27 grams of BCAAs will be administered twice-daily for 21 days
  Branched Chain Amino Acids: The three BCAAs will be combined together and dissolved in a flavored solution.
Period: Overall Study
Arm/Group | Placebo | Branched Chain Amino Acids (7.5g BID) | Branched Chain Amino Acids (15g BID) | Branched Chain Amino Acids (22.5g BID) | Branched Chain Amino Acids (27g BID)
Started | 8 | 8 | 9 | 9 | 8
Completed | 5 | 4 | 4 | 3 | 4
Not Completed | 3 | 4 | 5 | 6 | 4
Not completed — Lost to Follow-up | 3 | 4 | 1 | 6 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes all 42 patients randomized
Groups:
- Branched Chain Amino Acids (7.5g BID): 7.5 grams of BCAAs will be administered twice-daily for 21 days
  Branched Chain Amino Acids: The three BCAA's will be combined together and dissolved in a flavored solution.
- Branched Chain Amino Acids (22.5g BID): 22.5 grams of BCAAs will be administered twice-daily for 21 days
  Branched Chain Amino Acids: The three BCAA's will be combined together and dissolved in a flavored solution.
- Branched Chain Amino Acids (27g BID): 27 grams of BCAAs will be administered twice-daily for 21 days
  Branched Chain Amino Acids: The three BCAA's will be combined together and dissolved in a flavored solution.
- Total: Total of all reporting groups
Arm/Group | Placebo | Branched Chain Amino Acids (7.5g BID) | Branched Chain Amino Acids (15g BID) | Branched Chain Amino Acids (22.5g BID) | Branched Chain Amino Acids (27g BID) | Total
Number analyzed (Participants) | 8 | 8 | 9 | 9 | 8 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 7 | 9 | 9 | 6 | 37
  Between 18 and 65 years | 2 | 1 | 0 | 0 | 2 | 5
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 16.5 [14.5 to 18.5] | 15 [15 to 16.5] | 16 [14 to 17] | 15 [15 to 16] | 15.5 [13.5 to 21] | 15.5 [15 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 4 | 4 | 20
  Male | 4 | 4 | 5 | 5 | 4 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 3 | 0 | 1 | 5
  Not Hispanic or Latino | 7 | 8 | 6 | 9 | 7 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2 | 0 | 4
  White | 7 | 6 | 8 | 7 | 8 | 36
  More than one race | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 9 | 9 | 8 | 42
Days from injury to enrollment [Median (Inter-Quartile Range); unit: days] | 2 [1.5 to 2.5] | 2 [2 to 2.5] | 1 [0 to 2] | 2 [2 to 2] | 2 [1.5 to 3] | 2 [2 to 2.75]

OUTCOME MEASURES:

1. Primary Outcome: Reaction Time Difference Between Drug and Placebo Groups
Description: Processing speed subtest of the Axon Sports Computerized Cognitive Assessment Tool. The values provided are the median of log reaction time to the processing speed subtest, where a lower score indicates a faster time and thus improved processing speed.
Time Frame: Day 21
Population: Not all participants completed daily neurocognitive testing batteries, therefore there is incompleteness in the Day 21 values. In total, only 13 participants completed neurocognitive testing on day 21 (compared to 28 participants who completed full follow-up)
Measure: Median (Inter-Quartile Range); unit: log(milliseconds)
Groups:
- Branched Chain Amino Acids (15g BID): 15 grams of BCAAs will be administered twice-daily for 21 days
  Branched Chain Amino Acids: The three BCAAs will be combined together and dissolved in a flavored solution.
Arm/Group | Placebo | Branched Chain Amino Acids (7.5g BID) | Branched Chain Amino Acids (15g BID) | Branched Chain Amino Acids (22.5g BID) | Branched Chain Amino Acids (27g BID)
Number analyzed (Participants) | 4 | 1 | 2 | 2 | 4
log(milliseconds) | 2.44 [2.41 to 2.51] | 2.49 [2.44 to 2.55] | 2.52 [2.48 to 2.56] | 2.48 [2.46 to 2.57] | 2.48 [2.42 to 2.49]
Statistical Analysis 1: Comparison: Placebo vs Branched Chain Amino Acids (7.5g BID) vs Branched Chain Amino Acids (15g BID) vs Branched Chain Amino Acids (22.5g BID) vs Branched Chain Amino Acids (27g BID); Test type: Superiority; p = 0.871, Kruskal-Wallis

2. Secondary Outcome: Clinical Symptoms
Description: Evaluate whether BCAA supplementation reduces total symptom burden on a total symptom scale of 9 concussion symptoms rated each from 0-6, minimal value 0, maximum value 54, a higher score indicates a higher symptom burden and therefore a worse outcome
Time Frame: Day 21
Population: Only 20 of 38 subjects completed daily symptom and activity logs though the 3 weeks of the study
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Branched Chain Amino Acids (7.5g BID) | Branched Chain Amino Acids (15g BID) | Branched Chain Amino Acids (22.5g BID) | Branched Chain Amino Acids (27g BID)
Number analyzed (Participants) | 5 | 4 | 4 | 3 | 4
units on a scale | 3 [2 to 5] | 2 [0.5 to 3] | 0 [0 to 1.5] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Placebo vs Branched Chain Amino Acids (7.5g BID) vs Branched Chain Amino Acids (15g BID) vs Branched Chain Amino Acids (22.5g BID) vs Branched Chain Amino Acids (27g BID); Test type: Superiority; p = 0.140, Kruskal-Wallis

3. Secondary Outcome: Return to Physical Activity Baseline
Description: Determine whether BCAA supplementation more rapidly facilitates a return to physical baseline. The physical activity score is scaled on a 6 point Likert scale (0-5), where 0 represents no activity and 5 represents full activity, therefore a higher score represents a closer return to baseline activity by the end of the study period
Time Frame: Day 21
Population: Only 20 of 38 subjects completed daily symptom and activity logs though the 3 weeks of the study
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Branched Chain Amino Acids (7.5g BID) | Branched Chain Amino Acids (15g BID) | Branched Chain Amino Acids (22.5g BID) | Branched Chain Amino Acids (27g BID)
Number analyzed (Participants) | 5 | 4 | 4 | 3 | 4
score on a scale | 2 [1 to 2] | 1.5 [1 to 3] | 3 [1 to 5] | 3 [2 to 4] | 5 [3.5 to 5]
Statistical Analysis 1: Comparison: Placebo vs Branched Chain Amino Acids (7.5g BID) vs Branched Chain Amino Acids (15g BID) vs Branched Chain Amino Acids (22.5g BID) vs Branched Chain Amino Acids (27g BID); Test type: Superiority; p = 0.267, Kruskal-Wallis

4. Secondary Outcome: Neurocognitive Recovery-- Attention
Description: Determine whether administration of BCAAs improves the median log reaction time of the attention subtest of the neurocognitive testing battery. A lower median log reaction time represents improved attention
Time Frame: Day 21
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: log(milliseconds)
Arm/Group | Placebo | Branched Chain Amino Acids (7.5g BID) | Branched Chain Amino Acids (15g BID) | Branched Chain Amino Acids (22.5g BID) | Branched Chain Amino Acids (27g BID)
Number analyzed (Participants) | 4 | 1 | 2 | 2 | 4
log(milliseconds) | 2.65 [2.60 to 2.71] | 2.60 [2.55 to 2.65] | 2.73 [2.67 to 2.80] | 2.74 [2.62 to 2.86] | 2.69 [2.65 to 2.77]
Statistical Analysis 1: Comparison: Placebo vs Branched Chain Amino Acids (7.5g BID) vs Branched Chain Amino Acids (15g BID) vs Branched Chain Amino Acids (22.5g BID) vs Branched Chain Amino Acids (27g BID); Test type: Superiority; p = 0.476, Kruskal-Wallis

5. Secondary Outcome: Compliance and Adherence to Treatment
Description: Adherence to treatment among dosage groups, reported as the median percent drink consumed among the group across the study period, where 100% = all drink (2 doses per day x 21 days) consumed, and 0% represents no drink consumed
Time Frame: Day 21
Population: All 38 participants, minus the 4 who withdrew following randomization, are included in the adherence measure
Measure: Median (Inter-Quartile Range); unit: Percent of total drink consumed
Arm/Group | Placebo | Branched Chain Amino Acids (7.5g BID) | Branched Chain Amino Acids (15g BID) | Branched Chain Amino Acids (22.5g BID) | Branched Chain Amino Acids (27g BID)
Number analyzed (Participants) | 8 | 8 | 5 | 9 | 8
Percent of total drink consumed | 81 [14.3 to 87.9] | 64.3 [28.4 to 91.4] | 54.8 [15.0 to 55.6] | 23.8 [11.9 to 42.5] | 49.0 [22.7 to 72.6]
Statistical Analysis 1: Comparison: Placebo vs Branched Chain Amino Acids (7.5g BID) vs Branched Chain Amino Acids (15g BID) vs Branched Chain Amino Acids (22.5g BID) vs Branched Chain Amino Acids (27g BID); Test type: Superiority; p = 0.581, Kruskal-Wallis

6. Secondary Outcome: Tolerability of BCAA's Based on Adverse Events
Description: Assess the tolerability of BCAA doses based on subject reported adverse events, measured as the percent of participants in each study arm reporting adverse events
Time Frame: Day 21
Population: Adverse events were only evaluated for the 38 subjects who participated. The 4 subjects who withdrew did so prior to receiving any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Branched Chain Amino Acids (7.5g BID) | Branched Chain Amino Acids (15g BID) | Branched Chain Amino Acids (22.5g BID) | Branched Chain Amino Acids (27g BID)
Number analyzed (Participants) | 8 | 8 | 5 | 9 | 8
Participants | 3 | 3 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Placebo vs Branched Chain Amino Acids (7.5g BID) vs Branched Chain Amino Acids (15g BID) vs Branched Chain Amino Acids (22.5g BID) vs Branched Chain Amino Acids (27g BID); Test type: Superiority; p = 0.203, Fisher Exact

7. Secondary Outcome: Safety and BCAA Supplementation
Description: Asses the safety of BCAA doses in concussed athletes through subject reported serious adverse events (SAEs). Reported as the number of participants in each arm experiencing an SAE.
Time Frame: Day 21
Population: Only the 38 participants who received any study drug are included. The 4 who withdrew did so immediately after randomization before consuming any product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Branched Chain Amino Acids (7.5g BID) | Branched Chain Amino Acids (15g BID) | Branched Chain Amino Acids (22.5g BID) | Branched Chain Amino Acids (27g BID)
Number analyzed (Participants) | 8 | 8 | 5 | 9 | 8
Participants | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Branched Chain Amino Acids (7.5g BID) vs Branched Chain Amino Acids (15g BID) vs Branched Chain Amino Acids (22.5g BID) vs Branched Chain Amino Acids (27g BID); Test type: Superiority; p = 1.00, Fisher Exact

8. Secondary Outcome: Neurocognitive Recovery-- Working Memory
Description: Determine whether administration of BCAAs improves the the median of log reaction time of the working memory subtest of the neurocognitive testing battery. A lower median log reaction time represents improved working memory.
Time Frame: Day 21
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: log(milliseconds)
Arm/Group | Placebo | Branched Chain Amino Acids (7.5g BID) | Branched Chain Amino Acids (15g BID) | Branched Chain Amino Acids (22.5g BID) | Branched Chain Amino Acids (27g BID)
Number analyzed (Participants) | 4 | 1 | 2 | 2 | 4
log(milliseconds) | 2.69 [2.62 to 2.78] | 2.70 [2.59 to 2.80] | 2.84 [2.82 to 2.87] | 2.82 [2.68 to 2.97] | 2.74 [2.66 to 2.91]
Statistical Analysis 1: Comparison: Placebo vs Branched Chain Amino Acids (7.5g BID) vs Branched Chain Amino Acids (15g BID) vs Branched Chain Amino Acids (22.5g BID) vs Branched Chain Amino Acids (27g BID); Test type: Superiority; p = 0.482, Kruskal-Wallis

9. Secondary Outcome: Neurocognitive Recovery-- Visual Memory
Description: Determine whether administration of BCAAs improves the accuracy score of the visual memory subtest of the neurocognitive testing battery. A higher accuracy score (scaled 0-1.5) represents improved visual memory
Time Frame: Day 21
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Branched Chain Amino Acids (7.5g BID) | Branched Chain Amino Acids (15g BID) | Branched Chain Amino Acids (22.5g BID) | Branched Chain Amino Acids (27g BID)
Number analyzed (Participants) | 4 | 1 | 2 | 2 | 4
score on a scale | 1.24 [1.15 to 1.29] | 1.11 [0.88 to 1.34] | 0.99 [0.93 to 1.04] | 0.75 [0.22 to 1.27] | 1.05 [0.99 to 1.08]
Statistical Analysis 1: Comparison: Placebo vs Branched Chain Amino Acids (7.5g BID) vs Branched Chain Amino Acids (15g BID) vs Branched Chain Amino Acids (22.5g BID) vs Branched Chain Amino Acids (27g BID); Test type: Superiority; p = 0.393, Kruskal-Wallis

10. Secondary Outcome: Return to Baseline Cognitive Activity
Description: Determine whether BCAA supplementation more rapidly facilitates a return to cognitive activity baseline. The cognitive activity score is scaled on a 5 point Likert scale (0-4), where 0 represents no activity and 4 represents full activity, therefore a higher score represents a closer return to baseline cognitive activity by the end of the study period
Time Frame: Day 21
Population: Only 20 of 38 subjects completed daily symptom and activity logs though the 3 weeks of the study
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Branched Chain Amino Acids (7.5g BID) | Branched Chain Amino Acids (15g BID) | Branched Chain Amino Acids (22.5g BID) | Branched Chain Amino Acids (27g BID)
Number analyzed (Participants) | 5 | 4 | 4 | 3 | 4
score on a scale | 2 [2 to 4] | 3 [1.5 to 4] | 4 [3.5 to 4] | 4 [4 to 4] | 3 [1.5 to 4]
Statistical Analysis 1: Comparison: Placebo vs Branched Chain Amino Acids (7.5g BID) vs Branched Chain Amino Acids (15g BID) vs Branched Chain Amino Acids (22.5g BID) vs Branched Chain Amino Acids (27g BID); Test type: Superiority; p = 0.629, Kruskal-Wallis

11. Post Hoc Outcome: Regression Model Processing Speed Change
Description: Change in log reaction time of the neurocognitive testing processing speed score for increase of total study dose of 500 g in adjusted regression. This represents a change in the log reaction time for, on average, each increase of 500 g of study drug consumed between baseline and end of study period (between baseline, day 0, and day 21). A lower reaction time (on a scale of 2.35 to 2.80) indicates faster speed and thus improved neurocognitive function. The least squares mean for the model for each 500 g of drug consumed, with the standard error, are presented, as is the p-value for the slope parameter of the regression.
Time Frame: Baseline and 21 days
Population: 18 out of 38 participants completed at least 7 measurements of neurocognitive testing to contribute to the overall regression analysis. Participants across all treatment arms were combined for this regression as it was, rather than in intention-to-treat analysis, a dose response analysis testing the effect of actual study drug consumed
Measure: Least Squares Mean (Standard Error); unit: log(milliseconds)
Groups:
- Entire Study: Regression analysis was performed for all subjects with at least 7 reported measurements
Arm/Group | Entire Study
Number analyzed (Participants) | 18
log(milliseconds) | 0.008 (0.016)
Statistical Analysis 1: Comparison: Entire Study; Test type: Superiority; p = 0.624, Regression, Linear

12. Post Hoc Outcome: Regression Model Attention Change
Description: Change in log reaction time of the neurocognitive testing attention score for increase of total study dose of 500 g in adjusted regression. This represents a change in the log reaction time for, on average, each increase of 500 g of study drug consumed between baseline and end of study period (between baseline, day 0, and day 21). A lower reaction time (on a scale of 2.35 to 2.80) indicates faster speed and thus improved neurocognitive function. The least squares mean for the model for each 500 g of drug consumed, with the standard error, are presented, as is the p-value for the slope parameter of the regression.
Time Frame: Baseline and 21 days
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: log(milliseconds)
Groups:
- Entire Study: Regression analysis was performed for all subjects with at least 7 reported measurements of neurocognitive testing
Arm/Group | Entire Study
Number analyzed (Participants) | 18
log(milliseconds) | 0.014 (0.012)
Statistical Analysis 1: Comparison: Entire Study; Test type: Superiority; p = 0.2554, Regression, Linear

13. Post Hoc Outcome: Regression Model Working Memory Change
Description: Change in log reaction time of the neurocognitive testing working memory score for increase of total study dose of 500 g in adjusted regression. This represents a change in the log reaction time for, on average, each increase of 500 g of study drug consumed between baseline and end of study period (between baseline, day 0, and day 21). A lower reaction time (on a scale of 2.35 to 2.80) indicates faster speed and thus improved neurocognitive function. The least squares mean for the model for each 500 g of drug consumed, with the standard error, are presented, as is the p-value for the slope parameter of the regression.
Time Frame: Baseline and 21 days
Population: contribute to the overall regression analysis. Participants across all treatment arms were combined for this regression as it was, rather than in intention-to-treat analysis, a dose response analysis testing the effect of actual study drug consumed
Measure: Least Squares Mean (Standard Error); unit: log(milliseconds)
Arm/Group | Entire Study
Number analyzed (Participants) | 18
log(milliseconds) | 0.004 (0.0016)
Statistical Analysis 1: Comparison: Entire Study; Test type: Superiority; p = 0.7964, Regression, Linear

14. Post Hoc Outcome: Regression Mode Visual Learning Change
Description: Change in accuracy score of the neurocognitive testing processing speed score for increase of total study dose of 500 g in adjusted regression. This represents a change in the accuracy score for, on average, each increase of 500 g of study drug consumed between baseline and end of study period (between baseline, day 0, and day 21). The accuracy scale score is scaled from 0 to 1.5, and a higher score indicates higher accuracy and thus higher neurocognitive function. The least squares mean for the model for each 500 g of drug consumed, with the standard error, are presented, as is the p-value for the slope parameter of the regression.
Time Frame: Baseline and 21 days
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Entire Study
Number analyzed (Participants) | 18
score on a scale | -0.013 (0.046)
Statistical Analysis 1: Comparison: Entire Study; Test type: Superiority; p = 0.7749, Regression, Linear

15. Post Hoc Outcome: Total Symptom Score Change
Description: Change in total symptom score for increase of total study dose of 500 g in adjusted regression. This represents a change in the total symptom score for, on average, each increase of 500 g of study drug consumed between baseline and end of study period (between baseline, day 0, and day 21). The symptom score is scaled from 0-54, with a higher number representing a higher symptom burden and thus a worse outcome. The least squares mean for the model for each 500 g of drug consumed, with the standard error, are presented, as is the p-value for the slope parameter of the regression.
Time Frame: Baseline and 21 days
Population: 26 out of 38 participants completed at least 7 measurements of the daily symptom and activity questionnaire to contribute to the overall regression analysis. Participants across all treatment arms were combined for this regression as it was, rather than in intention-to-treat analysis, a dose response analysis testing the effect of actual study drug consumed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Entire Study, Symptom/Activity Questionnaire: Participants who completed at least 7 measurements of the daily symptom/activity questionnaire to contribute to the overall regression analysis
Arm/Group | Entire Study, Symptom/Activity Questionnaire
Number analyzed (Participants) | 26
score on a scale | -4.4 (1.4)
Statistical Analysis 1: Comparison: Entire Study, Symptom/Activity Questionnaire; Test type: Superiority; p = 0.0036, Regression, Linear

16. Post Hoc Outcome: Physical Activity Score Change
Description: Change in physical activity score for increase of total study dose of 500 g in adjusted regression. This represents a change in the physical activity score for, on average, each increase of 500 g of study drug consumed between baseline and end of study period (between baseline, day 0, and day 21). The physical activity scale is 0-5, with a maximum score of 5 representing full baseline physical activity. The least squares mean for the model for each 500 g of drug consumed, with the standard error, are presented, as is the p-value for the slope parameter of the regression.
Time Frame: Baseline and 21 days
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Entire Study, Symptom/Activity Questionnaire
Number analyzed (Participants) | 26
score on a scale | 0.503 (0.164)
Statistical Analysis 1: Comparison: Entire Study, Symptom/Activity Questionnaire; Test type: Superiority; p = 0.0053, Regression, Linear

17. Post Hoc Outcome: Regression Model Cognitive Activity Score Change
Description: Change in cognitive activity score for increase of total study dose of 500 g in adjusted regression. This represents a change in the cognitive activity score for, on average, each increase of 500 g of study drug consumed between baseline and end of study period (between baseline, day 0, and day 21). The cognitive activity scale is 0-4, with a maximum score of 4 representing full cognitive baseline activity. The least squares mean for the model for each 500 g of drug consumed, with the standard error, are presented, as is the p-value for the slope parameter of the regression.
Time Frame: Baseline and 21 days
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Entire Study, Symptom/Activity Questionnaire
Number analyzed (Participants) | 26
score on a scale | 0.051 (0.224)
Statistical Analysis 1: Comparison: Entire Study, Symptom/Activity Questionnaire; Test type: Superiority; p = 0.8234, Regression, Linear

ADVERSE EVENTS:
Time Frame: 21 days (duration of study period)
Arm/Group | Placebo | Branched Chain Amino Acids (7.5g BID) | Branched Chain Amino Acids (15g BID) | Branched Chain Amino Acids (22.5g BID) | Branched Chain Amino Acids (27g BID)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/9 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/9 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 3/8 | 3/8 | 1/9 | 0/9 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | Branched Chain Amino Acids (7.5g BID) (N=8) | Branched Chain Amino Acids (15g BID) (N=9) | Branched Chain Amino Acids (22.5g BID) (N=9) | Branched Chain Amino Acids (27g BID) (N=8)
Mild (not interfering with daily life) or Moderate (limitation to daily activity) (Gastrointestinal disorders) | 3 (5) | 3 (5) | 1 (1) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
There are several key limitations to our study that necessitate a larger, more definitive trial. Due to a combination of initially more strict inclusion criteria, and the impact of the coronavirus pandemic, our sample size was smaller than anticipated. This, combined with poorer than expected follow-up, led us to have to use alternative statistical analytic methods. We were further limited by missing data. This also necessitated the alternative analytic approach / post-hoc analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT01860404/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT01860404/ICF_001.pdf